CLINICAL TRIAL: NCT06563245
Title: A Phase II/III Study of Brentuximab Vedotin for Newly Diagnosed Classical Hodgkin Lymphoma in Chinese CAYA Based on PET/CT Assessment
Brief Title: Brentuximab Vedotin for Newly Diagnosed CHL in Chinese CAYA Based on PET/CT Assessment
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other); Najing Children's Hospital (Unknown); West China Second University Hospital (Other); Qilu Hospital of Shandong University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Tongji Hospital (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital of Anhui Medical University (Unknown); Children's Hospital of Hebei Province (Other); Children's Hospital of Henan Province (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-HL-2024
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Classical Hodgkin Lymphoma; Child; Adolescent; Young Adult; Metabolic Response; Survival; Treatment; Brentuximab Vedotin; PET Scan
MeSH Terms: interventions — Brentuximab Vedotin; Injections; Doxorubicin; Etoposide; Prednisone; Cyclophosphamide; Dacarbazine; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low risk group (Experimental): Stage IA , no bulky Stage IIA, no bulky
  Interventions: Drug: Brentuximab Vedotin for Injection; Radiation: response-adapted radiation; Drug: Doxorubicin; Drug: Etoposide; Drug: Prednisone; Drug: Cyclophosphamide
- Intermediate risk group (Experimental): Stage IA, with bulky Stage IIA, with bulky Stage IB, with/without bulky Stage IAE, with/without bulky Stage IIAE, with/without bulky Stage IIIA, with/without bulky
  Interventions: Drug: Brentuximab Vedotin for Injection; Radiation: response-adapted radiation; Drug: Doxorubicin; Drug: Etoposide; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Dacarbazine; Drug: Tislelizumab Injection; Drug: Bedamustine
- High risk group (Experimental): Stage IIB Stage IIIB Stage IV
  Interventions: Drug: Brentuximab Vedotin for Injection; Radiation: response-adapted radiation; Drug: Doxorubicin; Drug: Etoposide; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Dacarbazine; Drug: Tislelizumab Injection; Drug: Bedamustine

INTERVENTIONS:
Drug: Brentuximab Vedotin for Injection — 1.8mg/kg/dose (MAX 180 mg)
Radiation: response-adapted radiation — For patients who did not achieve complete metabolic response at early response assessment based on PET/CT result.
Drug: Doxorubicin — 25mg/m2/dose,
Drug: Etoposide — 125 mg/m2/dose
Drug: Prednisone — 20 mg/m2, BID, orally
Drug: Cyclophosphamide — 600 mg/m2/dose
Drug: Dacarbazine — 250 mg/m2/dose; For patients in intermediate/high risk group who did not achieve complete metabolic response at early assessment based on PET/CT results.
  Arms: High risk group; Intermediate risk group
Drug: Tislelizumab Injection — 3mg/kg/dose; For patients in intermediate/high risk group who did not achieve complete metabolic response at late assessment based on PET/CT results.
  Arms: High risk group; Intermediate risk group
Drug: Bedamustine — 180mg/m2/dose; For patients in intermediate/high risk group who did not achieve complete metabolic response at late assessment based on PET/CT results.
  Arms: High risk group; Intermediate risk group

SUMMARY:
Generally, pediatric patients tolerate acute toxicities but are vulnerable to late effects. Thus, increasing chemotherapy intensity to achieve more rapid complete early response to limit radiation therapy is worth testing. In this CCCG-HL-2024 study, Brentuximab vedotin (Bv) was used to replace VCR and bleomycin in the ABVE-PC regimen in the previous CCCG-HD-2018 study, respectively, to form a Bv-AEPC regimen for the treatment of newly diagnosed classic Hodgkin lymphoma (cHL) in children, adolescents and young adults. On the premise of maintaining a 4-year event free survival (EFS)>90% in the low-, intermediate-and high-risk groups, increase the early assessment complete response rate (the overall early complete response rate increased by 20%, that is, from 54.0% to 74.0%) to further reduce the proportion of children receiving radiotherapy to benefit them.

DETAILED DESCRIPTION:
In this CCCG-HL-2024 study, Brentuximab vedotin (Bv) was used to replace VCR and bleomycin in the ABVE-PC regimen in the previous CCCG-HD-2018 study, respectively, to form a Bv-AEPC regimen for the treatment of newly diagnosed classic Hodgkin lymphoma (cHL) in children, adolescents and young adults. Bv is currently the most widely used "new drug" in childhood cHL.

For patients in the intermediate/high-risk group who did not achieve metabolic complete remission rate (CMR) at the early assessment based on PET/CT results, an intensive regimen of Bv-Dac-APC (Bv-APC plus dacarbazine) was applied for 2 or 3 courses to further improve event-free survival without increasing long-term reproductive toxicity.

For patients in the intermediate/high-risk group who did not achieve CMR after the Bv-Dac-AEPC regimen, a modified Check Mate 744 regimen (PD-1 monoclonal antibody, Bv,+/-bedamostine, autologous stem cell transplantation/radiotherapy) was applied to improve the CMR of patients before irradiation, hoping to reduce the primary treatment failure rate to almost zero.

ELIGIBILITY:
Inclusion Criteria:

* Ages >=2~<35 years at the time of enrollment;
* Patients with newly diagnosed, pathologically confirmed classical Hodgkin lymphoma (HL) by at least 2 tertiary referral centers for pathology;
* Adequate organ function;
* Patients and/or their parents or legal guardians sign a written informed consent;

Exclusion Criteria:

* Patients with nodular lymphocyte-predominant HL;
* Patients with an immunodeficiency that existed prior to diagnosis; such as primary immunodeficiency syndromes, organ transplant recipients and children on current systemic immunosuppressive agents are not eligible;Patients known to be positive for HIV are not eligible.
* Patients who are pregnant; Lactating females who plan to breastfeed.
* Patients who received systemic corticosteroids within 28 days of enrollment on this protocol

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2029-11-15 (Estimated); Study Completion 2039-11-15 (Estimated)

PRIMARY OUTCOMES:
Early complete metabolic response rate for the entire group | 5 years
  Early complete metabolic response rate after 2 cycle of Bv-AEPC based on PET/CT result for the entire group
Late complete metabolic response rate in intermediate/high risk group | 5 years
  Late complete metabolic response rate based on PET/CT results for patients who did not achieve early complete metabolic response after 2 or 3 cycles of Bv-Dac-AEPC
Complete metabolic response rate in intermediate/high risk group after modified Check Mate 744 regimens | 5 years
  Complete metabolic response rate based on PET/CT results for patients who receive a modified Check Mate 744 regimen
Overall survival rate for the entire group and each risk group | 5 years
  the overall survival rate for all the patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: YI JIN GAO, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Monthly meeting within the group
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From October 15 2024 to the end of the study.
Access Criteria: After IRB approval is received.

REFERENCES:
- [Background] Huang J, Pang WS, Lok V, Zhang L, Lucero-Prisno DE 3rd, Xu W, Zheng ZJ, Elcarte E, Withers M, Wong MCS; NCD Global Health Research Group, Association of Pacific Rim Universities (APRU). Incidence, mortality, risk factors, and trends for Hodgkin lymphoma: a global data analysis. J Hematol Oncol. 2022 May 11;15(1):57. doi: 10.1186/s13045-022-01281-9. PMID 35546241
- [Background] Bao PP, Li K, Wu CX, Huang ZZ, Wang CF, Xiang YM, Peng P, Gong YM, Xiao XM, Zheng Y. [Recent incidences and trends of childhood malignant solid tumors in Shanghai, 2002-2010]. Zhonghua Er Ke Za Zhi. 2013 Apr;51(4):288-94. Chinese. PMID 23927803
- [Background] Nie DM, Yuan Q, Yu Y, Wu CJ, Guo X, Zhang AJ, Wang J, Xiao LY, Weng KZ, Fang YJ, Ju XL, Gao J, Xu ZJ, Yang LC, Liu AG, Gao YJ. [A multicenter study on childhood Hodgkin lymphoma treated with HL-2013 regimen in China]. Zhonghua Er Ke Za Zhi. 2022 Nov 2;60(11):1172-1177. doi: 10.3760/cma.j.cn112140-20220312-00196. Chinese. PMID 36319153
- [Background] Castellino SM, Pei Q, Parsons SK, Hodgson D, McCarten K, Horton T, Cho S, Wu Y, Punnett A, Dave H, Henderson TO, Hoppe BS, Charpentier AM, Keller FG, Kelly KM. Brentuximab Vedotin with Chemotherapy in Pediatric High-Risk Hodgkin's Lymphoma. N Engl J Med. 2022 Nov 3;387(18):1649-1660. doi: 10.1056/NEJMoa2206660. PMID 36322844
- [Background] Metzger ML, Link MP, Billett AL, Flerlage J, Lucas JT Jr, Mandrell BN, Ehrhardt MJ, Bhakta N, Yock TI, Friedmann AM, de Alarcon P, Luna-Fineman S, Larsen E, Kaste SC, Shulkin B, Lu Z, Li C, Hiniker SM, Donaldson SS, Hudson MM, Krasin MJ. Excellent Outcome for Pediatric Patients With High-Risk Hodgkin Lymphoma Treated With Brentuximab Vedotin and Risk-Adapted Residual Node Radiation. J Clin Oncol. 2021 Jul 10;39(20):2276-2283. doi: 10.1200/JCO.20.03286. Epub 2021 Apr 7. PMID 33826362
- [Background] Vardhana S, Cicero K, Velez MJ, Moskowitz CH. Strategies for Recognizing and Managing Immune-Mediated Adverse Events in the Treatment of Hodgkin Lymphoma with Checkpoint Inhibitors. Oncologist. 2019 Jan;24(1):86-95. doi: 10.1634/theoncologist.2018-0045. Epub 2018 Aug 6. PMID 30082490
- [Background] Harker-Murray P, Mauz-Korholz C, Leblanc T, Mascarin M, Michel G, Cooper S, Beishuizen A, Leger KJ, Amoroso L, Buffardi S, Rigaud C, Hoppe BS, Lisano J, Francis S, Sacchi M, Cole PD, Drachtman RA, Kelly KM, Daw S. Nivolumab and brentuximab vedotin with or without bendamustine for R/R Hodgkin lymphoma in children, adolescents, and young adults. Blood. 2023 Apr 27;141(17):2075-2084. doi: 10.1182/blood.2022017118. PMID 36564047
- [Background] Friedman DL, Chen L, Wolden S, Buxton A, McCarten K, FitzGerald TJ, Kessel S, De Alarcon PA, Chen AR, Kobrinsky N, Ehrlich P, Hutchison RE, Constine LS, Schwartz CL. Dose-intensive response-based chemotherapy and radiation therapy for children and adolescents with newly diagnosed intermediate-risk hodgkin lymphoma: a report from the Children's Oncology Group Study AHOD0031. J Clin Oncol. 2014 Nov 10;32(32):3651-8. doi: 10.1200/JCO.2013.52.5410. Epub 2014 Oct 13. PMID 25311218
- [Background] Kluge R, Kurch L, Georgi T, Metzger M. Current Role of FDG-PET in Pediatric Hodgkin's Lymphoma. Semin Nucl Med. 2017 May;47(3):242-257. doi: 10.1053/j.semnuclmed.2017.01.001. Epub 2017 Mar 6. PMID 28417854
- [Background] Mauz-Korholz C, Metzger ML, Kelly KM, Schwartz CL, Castellanos ME, Dieckmann K, Kluge R, Korholz D. Pediatric Hodgkin Lymphoma. J Clin Oncol. 2015 Sep 20;33(27):2975-85. doi: 10.1200/JCO.2014.59.4853. Epub 2015 Aug 24. PMID 26304892